CLINICAL TRIAL: NCT05227521
Title: The Feasibility of the Adapted H-GRASP Feedback Program for Perceived and Daily Life UL Activity in Patients With Good Observed But Low Perceived Activity in the Chronic Phase Post Stroke: a Pilot Study.
Brief Title: Feasibility of the Adapted H-GRASP Feedback Program in the Chronic Phase Post Stroke.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Prof Geert Verheyden, Professor, KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S66123; 1153320N (Other Grant/Funding Number: Research Foundation - Flanders (FWO))
Record Dates: First submitted 2022-01-14; First posted 2022-02-07 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Stroke
Keywords: upper limb; daily life activity; home-based exercise program; feedback; perceived activity
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- AH-GRASP feedback intervention group (Experimental): All study participants will receive the AH-GRASP feedback intervention.
  Interventions: Behavioral: Adapted H-GRASP feedback program

INTERVENTIONS:
Behavioral: Adapted H-GRASP feedback program — Combination of the Home-Graded Repetitive Arm Supplementary Program with in home accelerometer-based feedback

SUMMARY:
In a recent cross-sectional study, it was shown that people with a good observed upper limb (UL) motor function but low perceived UL activity show a reduced daily-life UL activity. The investigators will now investigate the feasibility of a phone-monitored home exercise and feedback program for the UL following stroke and the preliminary effects on the perceived UL activity and actual daily-life UL activity for participants with good observed UL motor function but low perceived UL activity in the chronic phase post-stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written informed consent of the participant has been obtained prior to any screening procedures
2. First-ever unilateral, supratentorial stroke, as defined by the American Heart Association/American Stroke Association
3. Minimum six months after stroke
4. Living in the community
5. ≥18 years old
6. Good observed UL motor function but low perceived UL activity. Good observed UL motor function is defined as a score >50/66 on the Fugl-Meyer Assessment-Upper Extremity (FMA-UE). Low perceived UL activity is defined as a score ≤75/100 on the hand subscale of the Stroke Impact Scale version 3.0 (SIS-Hand).

Exclusion Criteria:

1. Other neurological condition than stroke
2. Musculoskeletal disorder that affects UL use
3. No informed consent
4. Participation in an interventional Study with an investigational medicinal product (IMP) or device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2023-06-25 (Actual); Study Completion 2023-06-25 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 45 days (post-intervention)
  % of individuals who were eligible and agreed to participate
Retention rate | 45 days (post-intervention)
  % of participants who completed the intervention
Adherence to the intervention protocol | 45 days (post-intervention)
  % of participants who achieved 12 hours of average weekly exercise
Safety | 45 days (post-intervention)
  # of participants with increased pain while performing exercises as measured by visual analogue scale
Activity ratio | Day 1 (enrolment)
  Contribution to the activity of one upper limb (UL) versus the other: hours of activity of the affected divided by the unaffected UL
Activity ratio | Day 17 (baseline)
  Contribution to the activity of one upper limb (UL) versus the other: hours of activity of the affected divided by the unaffected UL
Activity ratio | 45 days (post-intervention)
  Contribution to the activity of one upper limb (UL) versus the other: hours of activity of the affected divided by the unaffected UL
Hand subscale of the Stroke Impact Scale version 3.0 (SIS-Hand) | Day 1 (enrolment)
  Perceived activity of the affected UL. Minimum 0 - maximum 100; higher scores mean better outcome.
Hand subscale of the Stroke Impact Scale version 3.0 (SIS-Hand) | Day 17 (baseline)
  Perceived activity of the affected UL. Minimum 0 - maximum 100; higher scores mean better outcome.
Hand subscale of the Stroke Impact Scale version 3.0 (SIS-Hand) | 45 days (post-intervention)
  Perceived activity of the affected UL. Minimum 0 - maximum 100; higher scores mean better outcome.

SECONDARY OUTCOMES:
Fugl-Meyer motor assessment - upper extremity (FMA-UE) | Day 1 (enrolment), day 17 (baseline), 45 days (post-intervention)
  Observed motor function of the affected UL (shoulder, arm, wrist, hand, and fingers)
Action Research Arm Test (ARAT) | Day 17 (baseline), 45 days (post-intervention)
  Grasp, grip, pinch and gross movement of the affected UL
Motor Activity Log - 14 Item Version Amount Of Use (MAL-14 AOU) | Day 17 (baseline), 45 days (post-intervention)
  Patient-reported amount of UL use in daily life
Motor Activity Log - 14 Item Version Quality Of Movement (MAL-14 QOM) | Day 17 (baseline), 45 days (post-intervention)
  Patient-reported quality of UL use in daily life
Erasmus modified Nottingham Sensory Assessment (Em-NSA) | Day 17 (baseline), 45 days (post-intervention)
  Sensory assessment of the UL
simplified modified Rankin Scale questionnaire (smRSq) | Day 17 (baseline), 45 days (post-intervention)
  Global disability. Minimum 0 - maximum 5; higher scores mean worse outcome.
Hospital Anxiety and Depression Scale (HADS) | Day 17 (baseline), 45 days (post-intervention)
  Symptoms of anxiety and depression. Minimum 0 - maximum 42; higher scores mean worse outcome.
Confidence in Arm and Hand Movement Scale (CAHM) | Day 17 (baseline), 45 days (post-intervention)
  Perceived self-efficacy in performing tasks with the affected UL. Minimum 0 - maximum 100; higher scores mean better outcome.
Visual Analogue Scale (VAS) | Day 17 (baseline), 45 days (post-intervention)
  Pain intensity in the affected UL from 0 (no pain) to 10 (extreme). Minimum 0, maximum 10, higher scores mean worse outcome.
EuroQol Five Dimensions Five Levels Questionnaire (EQ-5D-5L) | Day 17 (baseline), 45 days (post-intervention)
  Health-related quality of life. Minimum 0, maximum 100, higher scores mean better outcome.
Hours of UL activity | Day 1 (enrolment), day 17 (baseline), 45 days (post-intervention)
  Sum of all seconds recorded when the activity count was nonzero and converted to hours
Bilateral magnitude | Day 1 (enrolment), day 17 (baseline), 45 days (post-intervention)
  Intensity of the movement: sum of the vector magnitude from the two ULs
Magnitude ratio | Day 1 (enrolment), day 17 (baseline), 45 days (post-intervention)
  Contribution to the activity of one limb versus the other: natural log of the vector magnitude of the affected UL divided by the vector magnitude of the unaffected UL, whereby values greater than and less than -7 were replaced by 7 and -7, respectively, to categorize single limb movement.
Density plot | Day 1 (enrolment), day 17 (baseline), 45 days (post-intervention)
  Graphical representation of accelerometry data from both ULs

OTHER OUTCOMES:
Demographics | Day 1 (enrolment)
  Participant demography
Stroke event data | Day 1 (enrolment)
  Disease characteristics
National Institutes of Health Stroke Scale (NIHSS) | Day 1 (enrolment)
  Neurological impairments. Minimum 0, maximum 42, higher scores mean worse outcome.
Edinburgh Handedness Inventory (EHI) | Day 1 (enrolment)
  Handedness
Montreal Cognitive Assessment (MoCA) | Day 1 (enrolment)
  Cognitive function
Apples Test | Day 1 (enrolment)
  Visuospatial neglect
Barthel Index (BI) | Day 1 (enrolment)
  Performance in activities of daily living

CONTACTS AND LOCATIONS:
Overall Officials: Geert Verheyden, Professor, Principal Investigator — KU Leuven
Locations (1):
- Private physiotherapy practices, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No